CLINICAL TRIAL: NCT04008888
Title: Phase II Open Lable Clinical Study Efficacy and Safety of the Holistic Treatment for Young Patients With High-Risk Multiple Myeloma
Brief Title: a Clinical Trial of Efficacy and Safety of the Holistic Treatment of Young High-risk Multiple Myeloma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Qiu Lugui, Chief physician, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IHBDH-IIT2016011
Record Dates: First submitted 2019-06-21; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Multiple Myeloma; Plasma Cell Leukemia; Extramedullary Plasmacytoma; Loss of Chromosome 17p; t(14;16); t(4;14); T(14;20); 1Q21 Amplification; Complex Karyotype
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell; Chromosome 17 deletion | interventions — Melphalan; fludarabine; fludarabine phosphate; Dexamethasone; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A:Allogeneic Stem Cell Transplant Group (Experimental): Fludarabine+Melphalan followed by Allogeneic SCT.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Melphalan Given IV; Drug: Fludarabine Injection; Drug: PI and dexamethasone as maintenance therapy
- B:Autologous Stem Cell Transplant (Experimental): Melphalan followed by Autologous SCT.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation x 1 or x 2; Drug: Melphalan Given IV; Drug: PI and dexamethasone as maintenance therapy
- C:Non-Transplant (Experimental): Consolidated Chemotherapy for Patients Unable to Receive Transplantation
  Interventions: Drug: PI and dexamethasone as maintenance therapy; Drug: PI+IMids+Dexamethasone as Consolidated Chemotherapy

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Allogeneic Stem Cell Transplant: Day 0 Infusion of allogeneic peripheral blood stem cells. For the allogeneic matched-related donors peripheral blood stem cells will be harvested with GCSF mobilization and infused fresh to the recipients.
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HCT; SCT
  Arms: A:Allogeneic Stem Cell Transplant Group
Procedure: Autologous Hematopoietic Stem Cell Transplantation x 1 or x 2 — Autologous hematopoietic stem cell transplantation :Stem cell mobilization with granulocyte colony-stimulating factor (GCSF) at a dose of 10 μg/kg/day followed collecting CD34+ peripheral blood stem cells . Day 0 Infusion of autologous stem cells. Patients during 3-6 months after the 1st SCT will undergo a 2nd SCT. Patients who had not enough PBSC will undergo a 1st SCT.
  Other Names: autologous stem cell transplantation
  Arms: B:Autologous Stem Cell Transplant
Drug: Melphalan Given IV — conditioning regimen: autologous ARM: Day -2 Melphalan 200 mg/m^2/day IV over 30 minutes. allogeneic ARM: Day -4, Day -3 Melphalan 70 mg/m^2/day IV over 30 minutes
  Other Names: Alkeran
  Arms: A:Allogeneic Stem Cell Transplant Group; B:Autologous Stem Cell Transplant
Drug: Fludarabine Injection — conditioning regimen:Days -6,-5,-4,-3 Fludarabine 30 mg/m^2/day IV
  Other Names: Fludara
  Arms: A:Allogeneic Stem Cell Transplant Group
Drug: PI and dexamethasone as maintenance therapy — Bortezomib and dexamethasone(VD),Ixazomib and dexamethasone(ID)
  Other Names: VD; ID
Drug: PI+IMids+Dexamethasone as Consolidated Chemotherapy — Oral lenalidomide at the starting dose of 25mg on days 1-21 every 28 days or days 1-14 every 21 days. Dexamethasone at 20mg twice weekly on days 1,2,4,5,8,9,11&12 of each 21-day.
  Other Names: VRD; IRD; VDPACE; VDECP
  Arms: C:Non-Transplant

SUMMARY:
The clinical trial was conducted in a cohort of young, high-risk myeloma patients who were designed to receive a combination of high-dose chemotherapy with allogeneic or autologous hematopoietic stem cell transplantation. The objective was to assess the progression free survival (PFS), overall survival (OS),and overall response rate (ORR) of the overall treatment.

DETAILED DESCRIPTION:
50 cases of HR-NDMM patients were divided into two groups nonrandomizedly. TE group received hematopoietic stem cell transplantation after induction therapy. Allo-sct for the young patients with suitable donors, Asct for the others. TNE group received consolidation therapy after induction therapy. All patients received PI-based maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of high-risk multiple myeloma

   In addition, patients must meet at least one of the following criteria I-IX (I-VIII at time of diagnosis or pre-autograft):

   I.Complex karyotype

   II.Fluorescent in situ hybridization (FISH) translocation 4:14 or 14:16,

   III.FISH translocation 1q21,

   IV.FISH deletion 17p,

   V.R-ISS III stage,

   VI.Two or more high-risk cytogenetic abnormalities exist

   VII.Plasma cell leukemia

   VIII.Extramedullary plasmacytoma

   IX.Recurrent or non-responsive (less than partial remission [PR]) MM after at least 4 cycles of PI/IMids-based chemotherapy
2. candidate for high-dose chemotherapy with stem cell transplantation
3. ECOG performance status score of 0,1,or2 -

Exclusion Criteria:

1. The current diagnosis of smoldering multiple myeloma, monoclonal gammopathy of undetermined significance of disease, Waldenstr o m macroglobulinemia.
2. during the first 5 years of the study, there were no other malignancies, including basal cell carcinoma or in situ cervical cancer.
3. according to the National Cancer Institute general toxicity criteria (NCI CTC), subjects had peripheral neuropathy of grade 2 or above:
4. were enrolled within 6 months before had a myocardial infarction, or New York Heart Association (NYHA) III or IV heart failure ,uncontrolled angina, uncontrolled severe ventricular arrhythmias or ECG evidence of acute ischemia or conduction system abnormalities and activity the clinical significance of pericardial disease, or cardiac amyloidosis -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival(PFS) | 1 Year post-autograft
  PFS is defined as the duration from the data of registration to either progressive disease or death, whichever comes first.

SECONDARY OUTCOMES:
overall response(ORR) | 1 Year post-autograft
  ORR is defined as the proportion of subjects who achieve PR to better rate, according to the IMWG criteria
overall survival(OS) | 1 Year post-autograft
  OS is defined as the duration from the data of registration to death.If the subject is alive, the data will be censored as being alive; the vital status is unknown as last known.
Number of Patients With Grade II-IV Acute Graft-versus-Host-Disease and/or Chronic Extensive Graft-versus-Host-Disease | 1 year post-allograft
  aGVHD The diagnosis of aGVHD is identified through various stages and grading of the disease related to Skin (Rash), Gut (Diarrhea, Nausea/vomiting and/or anorexia) and the liver (Bilirubin) assessed by severity and grading scale outlined in the section Grafts vs Hosts by Sullivan (1999).
  GVHD Grades Grade I: 1-2 Skin Rash; No gut or liver involvement Grade II: Stage 1-3 Skin rash; Stage 1 gut and/or stage 1 liver involvement Grade III: Stage 2-4 gut involvement and/or stage 2-4 liver involvement with or without rash Grade IV: Pattern and severity of GVHD similar to grade 3 with extreme constitutional symptoms or death cGVHD The diagnosis of cGVHD requires at least one manifestation that is distinctive for chronic GVHD as opposed to acute GVHD. In all cases, infection and others causes must be ruled out in the differential diagnosis of chronic GVHD.
Non-relapse Mortality (NRM) | 1 year post-allograft
  Number of patients with non-relapse mortalities
Number of Patients Who Had Infections | 1 Year post-autograft
  Number of patients who had infections

CONTACTS AND LOCATIONS:
Overall Officials: Lu G Qiu, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No